CLINICAL TRIAL: NCT01794897
Title: Valacyclovir Augmentation for Cognitive and Functional Remediation in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Dr. Ram Manohar Lohia Hospital (Other Government); Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor of Psychiatry and Human Genetics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRO11120013
Record Dates: First submitted 2013-02-06; First posted 2013-02-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Herpes Simplex; Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Herpes Simplex; Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valacyclovir treatment (Experimental): Drug: Experimental: Valacyclovir treatment. Patients will have a placebo run-in for two weeks after which they will be evaluated for the variables of interest and then randomized to either Valacyclovir (VAV) or placebo (PLA) group in a 1:1 proportion. The VAV group will receive 1.5 g Valacyclovir by mouth, twice daily for 16 weeks, after which they will be followed up without VAV for 4 weeks to monitor delayed adverse effects.
  Interventions: Drug: Experimental: Valacyclovir treatment; Drug: Placebo comparator
- Placebo (Placebo Comparator): Placebo comparator: Patients will have a placebo run-in for two weeks after which they will be evaluated for the variables of interest and then randomized to either VAV or placebo group in a 1:1 proportion. Subjects in the placebo arm will receive placebo for 16 weeks, after which they will be followed up without placebo for 4 weeks to monitor delayed adverse effects.
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Experimental: Valacyclovir treatment — Patients will have a placebo run-in for two weeks after which they will be evaluated for the variables of interest and then randomized to either VAV or placebo group in a 1:1 proportion. The VAV group will receive 1.5 g Valacyclovir by mouth, twice daily for 16 weeks, after which they will be followed up without VAV for 4 weeks to monitor delayed adverse effects.
  Arms: Valacyclovir treatment
Drug: Placebo comparator — Patients will have a placebo run-in for two weeks after which they will be evaluated for the variables of interest and then randomized to either VAV or placebo group in a 1:1 proportion. Subjects in the placebo arm will receive placebo for 16 weeks, after which they will be followed up without placebo for 4 weeks to monitor delayed adverse effects.

SUMMARY:
The effects of Valacyclovir (VAV) augmentation or placebo (PLA) as adjuncts to conventional antipsychotic drug treatment will be evaluated among patients with schizophrenia who have been exposed to herpes simplex virus type 1 (HSV-1). Hypothesis: Valacyclovir (VAV) augmentation improves (a) cognitive and (b) overall function among Herpes Simples Virus 1 (HSV-1) exposed early course schizophrenia patients.

DETAILED DESCRIPTION:
Design: We propose a randomized double blind placebo controlled study of patients with early course Schizophrenia (SZ) / schizoaffective disorder (SZA) patients exposed to HSV-1, who are receiving antipsychotic drugs. The effects of VAV augmentation or PLA as adjuncts to conventional antipsychotic drug treatment will be evaluated. As outcomes, we will evaluate clinical symptoms, cognitive variables, overall function (including social function) and side effects. The participants will be under the direct care of the Indian investigators during the study. Ratings will be performed blind by research staff. We will pre-screen for HSV-1 exposure. There will be a 2 week placebo run in phase, 16 week augmentation and 4 week follow up to identify post-treatment side effects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Both genders, ages 18-50 years
* Schizophrenia / schizoaffective disorder (DSM IV).
* Stable dose of antipsychotic for > 1 month, continued throughout the study.
* Score 4 or more on one or more items of the Positive and Negative Syndrome Scale.
* Exposed to HSV-1: serum antibody assays.

Exclusion Criteria:

* Substance abuse in the past month/dependence past 6 months.
* History / current medical /neurological illnesses e.g., epilepsy.
* Pregnancy.
* History of immune disorders, HIV infection, or receiving immune-suppressants.
* Receiving regular antiviral therapy.
* History of hypersensitivity to Valacyclovir.
* Mental retardation as defined in DSM IV.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2013-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cognition | Assessed at week 16
  The following measures will be used to assess cognitive functioning both before and after treatment with Valacyclovir:
  Cognition: (1) Trail Making Test (TMT). This paper and pencil test is a convenient estimate of cognitive function, principally focusing on attention, working memory and executive function. (2) Computerized Neuropsychological Battery (CNB). We have validated a Hindi version of the Penn CNB and administered it to over 300 Indian participants. The CNB includes cognitive measures that distinguish SZ cases and relatives from controls. Accuracy and response time are recorded. Cognitive domains assessed: Abstraction and mental flexibility; Attention; Verbal Memory; Face Memory; Spatial Memory; Spatial Processing; Sensory-motor Dexterity; Emotion Processing.

SECONDARY OUTCOMES:
Clinical Severity | Assessed at week 16
  Clinical Severity will be measured by the following assessments: (i) Positive and Negative Syndrome Scale (PANSS. The PANSS is 7 point rating scale for 30 psychopathological items based on interviews or reports. (ii) Clinical Global Impression - Severity (CGI-S). The CGI-S is a 7-point scale that rates the severity of the patient's illness at the time of assessment.
Social Function | Assessed at week 16
  Social function will be measured by: (1) Independent Living Skills Survey (ILSS), a comprehensive, validated measure of functional living skills including self rated and observer rated portions (2) Sheehan's disability scale (SDS), a self-report tool that assesses functional impairment in work/school, social and family life with a 10-point visual analogue scale; (3) Global Assessment of Function (GAF), a global measure of function and symptom severity (4) Quality of Life Scale (QOL) measures interpersonal, social and occupational functioning.
Side Effects | Assessed at week 16
  Side effects will be assessed using: (1) Abnormal Involuntary Movement Scale This scale rates the severity of dyskinetic movements. Orofacial, neck-trunk and distal (limb) movements are rated separately. 2) Barnes Akathisia Scale: A rating scale to assess the severity of drug-induced akathisia.

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit Nimgaonkar, MD, PhD, Principal Investigator — University of Pittsburgh; Smita Deshpande, MD, Principal Investigator — Dr. Ram Manohar Lohia Hospital
Locations (1):
- Dr. Ram Manohar Lohia Hospital, Delhi, India